CLINICAL TRIAL: NCT02798588
Title: Improving Awakening Prognostication After Non Anoxic Coma Using PET-MRI in Intensive Care Unit
Acronym: ETIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL15_0669; 2015-A01886-43 (Other: ID-RCB)
Record Dates: First submitted 2016-05-27; First posted 2016-06-14 (Estimated); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: Coma
Keywords: coma; prognosis; comparative study; functional imaging; PET-MRI; electrophysiology
MeSH Terms: conditions — Coma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Comatose patients in ICU (Experimental)
  Interventions: Radiation: PET-MRI

INTERVENTIONS:
Radiation: PET-MRI — 18Fluoro-Desoxy-Glucose's infusion for PET (glucose neural metabolism assessment, with quantitative information permitted by radioactivity monitoring through arterial catheter ; dosage = 1,5 MBq/Kg + 18,5 MBq as loading dose 5 min= Outside the scanner, Installation and movement management: Curare+/- sedative injection with standardized routine care protocol 10 min= Outside the scanner, Starting PET continuous acquisitionT= 0, Morphological MRI sequences- 3DT1, 3DFlair, T2SE, T2 HR on brainstem, Susceptibility and simple Diffusion Weighted Imaging-Specifically dedicated MR sequences based upon clinical issues 25 min, MRI in Resting state N°1 (global short-term functional connectivity)13 min, MRI DTI acquisition, 64 directions, sensitive to white matter injury 8 min, IRM in 2D-Arterial Spin Labelling:Quantitative Cerebral blood flow information (no Gadolinium)->8 min, IRM in Resting state 2 (repeated occurrence to assess stationarity) 13 min, End of PET continuous acquisition

SUMMARY:
In last decades, several advances in the neuro-intensive management have lead to decrease mortality in Intensive Care Units. A significant morbidity remains as patients survive after a traumatic coma with uncertain quality of awakening and a high risk of functional disability. Predicting awareness recovery and functional disability of those who will awake constitutes a major challenge to inform patients' relatives, to give the best chances in terms of rehabilitation resources or to adapt intensive cares to a reasonable level. Tools currently available are not sufficient neither to predict bad awakening outcome nor to predict good functional outcome. In many countries, life's support cessation is a constant call for robust evaluation as soon as possible in ICU but it is mandatory to reach a positive predictive value of non-awaking close to 100%. Many clinical, electro-physiological, biological, radiological and functional parameters have been conducted with comatose patients assuming the purpose to predict outcome. Regarding unfavourable outcome, the gold standard is the abolition of the N20 component of somatosensory evoked potentials but the specificity is high enough only for patients with anoxic coma. Several neurophysiological markers such as MMN, P300 are correlated to a favourable outcome but the sensitivity and specificity remains low for patients who suffered a severe traumatic brain injury. New Diffusion Tensor imaging sequences provide complementary information to detect small structural lesions (diffuse axonal lesions). Recently, functional MRI analyzing Resting State has also been proposed as a prognostic marker during coma. PET using Fluoro-Desoxy-Glucose is able to assess the metabolism in key regions of the awakening network in either anaesthesia or sleep. Recent studies have reported interesting results at the chronic stage but to knowledge, these tools have only been used to address pathophysiology's issues and never to improve coma prognosis at the initial stage. The investigators hypothesize that the heterogeneity of the population requires a global and accurate assessment of the central nervous system, combining structural, metabolic and functional information in order to refine the prognosis.

The protocol integrates in one-sequence most radiological markers of brain injury within a unique PET-MRI in Lyon. The most relevant originality of the study consists in confronting FDG-PET and MRI sequences to a large clinical, electrophysiological and biological battery. The added clinical value would be to question the synergistic effect of each parameter and to find out which ones are the most useful for awakening prediction, as they have not been compared in a multi-parametric database.

PET-MRI, as a new device combining physiological and prognostic questioning, allows us:

* to implement a more integrative physio-pathological analysis
* to avoid the cofounding effect of awareness' fluctuations in recording simultaneously multiple functional imaging techniques.

The RS will be analyzed at 2 epochs in order to assess the stability of brain connectivity, related to neuronal activity (glucose metabolism) and brain perfusion.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting either vascular or traumatic lesions
2. Patients with no response to simple command 48h after sedation's cessation
3. Patients included between 7 days (to reduce the effect of early oedema) and 30 days after the coma (to control the homogeneity of our cohort)
4. Patients included between 18 and 75 years old, to limit the risk of care withdrawal for poor previous medical condition
5. Patients evaluated by a global electrophysiological assessment at beside in ICU in a short delay before or after PET-MRI

Exclusion Criteria:

1. Patient with an associated anoxic encephalopathy
2. Patients with contra-indication to MRI
3. Patients with hypersensibility to the active molecules (FDG) or to one of this excipient
4. Pregnant women
5. Minor patients
6. Patients under legal protection
7. Patients not affiliated to French health care system
8. Patients in poor medical condition (hemodynamic, respiratory instability)
9. Patients moribund or with previous decision of care withdrawal
10. Absence of relatives to give written consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2020-06-04 (Actual); Study Completion 2020-06-04 (Actual)

PRIMARY OUTCOMES:
Analysis of feasibility (pilot study) with Number of patients included during a 12-months period | at 12 months
Analysis of feasibility (pilot study) with ratio of patient included vs patient admissible according to the screening | at 12 months
Analysis of feasibility (pilot study) with respect of deadline for completion of PET MRI | at 12 months
Analysis of security (pilot study) with tolerance of the PET-MRI | at 12 months

SECONDARY OUTCOMES:
Unfavorable clinical evolution towards awareness (dichotomic criteria : absence of awareness with functional communication) | at 12 month
  Building a prognostic tool including miscellaneous parameters (clinical, biological, electrophysiological, metabolic PET and multimodal MRI) for the prediction of an unfavourable outcome (death, vegetative state, minimally conscious state) at 1 year after a non-anoxic brain injury (focal or multifocal; either traumatic or vascular causes)
Unfavorable clinical evolution in absence of awareness (ordinal criteria within unfavorable outcome) with Coma Recovery Scale-Revised | at 12 month
  Defining an association of criteria, which are available in the 1st month after coma, that are able to predict at 1 year with a high positive predictive value the level of disorder of consciousness in the subgroup with unfavourable outcome in analyzing (according to Coma Recovery Scale-Revised) the evolution of :
  * vegetative state patients
  * minimally-conscious patients
  * dead patients
Functional clinical evolution in presence of awareness (ordinal criteria within favorable outcome) according to Glasgow Outcome Scale (GOS) | at 12 month
  Defining an association of criteria which are available in the 1st month after coma, that are able to predict at 1 year with a high positive predictive value the quality of functional outcome in the subgroup with favourable outcome in analyzing the level of autonomy according to Glasgow Outcome Scale (GOS)

CONTACTS AND LOCATIONS:
Overall Officials: Florent GOBERT, MD, Principal Investigator — Réanimation polyvalente neurologique Hospices Civils de Lyon
Locations (1):
- Réanimation polyvalente neurologique Hôpital Neurologique HCL, Bron, France

IPD SHARING:
Plan to Share IPD: No